CLINICAL TRIAL: NCT02392819
Title: Food Design for Improved Cognitive Performance
Brief Title: Effects on Metabolism and Cognitive Functions of a Commonly Used Commercial Food Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Anne Nilsson, PhD, Associate Professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LundU
Record Dates: First submitted 2015-03-02; First posted 2015-03-19 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Postprandial Blood Glucose Regulation
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- test product (Experimental): Arm: Panax ginseng
  Interventions: Dietary Supplement: Panax ginseng
- placebo product (Placebo Comparator): Arm: a placebo with similar appearance but without Panax ginseng. The tablet include all the other non-active bulk ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Panax ginseng — Pananx ginseng is provided prior to a standardised breakfast, effects on test variables are determined at fasting and repeatedly postprandially the breakfast
  Arms: test product
Dietary Supplement: Placebo
  Arms: placebo product

SUMMARY:
This project evaluate effects of a commonly used food supplement on glucose metabolism and cognitive function.

DETAILED DESCRIPTION:
The test product has previously been suggested to elicit beneficial effects on glucose metabolism and cognitive performance. The purpose with this study is to evaluate metabolic effects and effects on mood variables of the test product provided at breakfast. Test variables are determined at fating and postprandial a standardised breakfast. The results are compared with effects after a placebo product.

ELIGIBILITY:
Inclusion Criteria:

* age between 40-60 years, normal BMI, healthy, non-smokers

Exclusion Criteria:

* metabolic disorders or gastro- intestinal disease, intake of probiotics- or antibiotics during the last 2 weeks prior to the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
blood glucose | 4 hours
  capillary blood glucose concentrations are determined at fasting and then repeatedly after a standardised breakfast

SECONDARY OUTCOMES:
serum insulin | 4 hours
  capillary serum insulin concentrations are determined at fasting and then repeatedly after a standardised breakfast
Mood as measured by ratings on 100 mm visual analog scales( VAS rating scales) | 4 hours
  measures of 6 mood variables (sad-glad, depressed-happy, displeased-pleased, dull-peppy, passive-Active, sleepy-awake) repeatedly in the postprandial period after breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Nilsson, PhD, Principal Investigator — Food for Health science Centre
Locations (1):
- Food for Health Science Centre, Medicon Village, Lund, Sweden